CLINICAL TRIAL: NCT05782751
Title: Growth Factor Enhanced Matrix Combined Either With Free Connective Tissue Graft or With Collagen Membrane in the Treatment of Miller Class II Gingival Recession
Brief Title: Growth Factor Enhanced Matrix With Subepithelial Connective Tissue Graft or Collagen Membrane in Treatment of Gingival Recession
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, malak mohamed shoukheba, professor of oral medicine, oral periodontology, oral diagnosis and diagnosis, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 6
Record Dates: First submitted 2023-02-27; First posted 2023-03-24 (Actual); Last update posted 2023-03-24 (Actual); Status verified 2023-03

CONDITIONS: GINGIVAL RECESSION
Keywords: Gingival recession; free subepithelial connective tissue graft; collagen membrane; growth factor enhanced matrix 21 s
MeSH Terms: conditions — Gingival Recession

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- (groupI) (Experimental): 10 recession sites treated by (GEM 21s) ® with free connective tissue graft
  Interventions: Procedure: GROUPI
- (groupII) (Active Comparator): 10 recession sites GEM 21s with collagen membrane
  Interventions: Procedure: GROUP II

INTERVENTIONS:
Procedure: GROUPI — 10 sites treated with Free connective tissue graft (FCTG) + growth factors enhanced matrix 21 s GEM 21S + coronally advanced flap (CAF)
  Other Names: free connective tissue graft; growth factors enhanced matrix 21s (GEM21s); coronally advanced flap
  Arms: (groupI)
Procedure: GROUP II — 10 sites treated withCollagen membrane + GEM 21S + coronally advanced flap (CAF)
  Other Names: collagen membrane; coronally advanced flap
  Arms: (groupII)

SUMMARY:
The study aimed to compare, the effectiveness of Growth Factor Enhanced Matrix (GEM 21s) ® combined either with free connective tissue graft or collagen membrane in the treatment of Miller class II gingival recession.

DETAILED DESCRIPTION:
Materials and Methods: Twenty sites in 10 patients, with class II Miller gingival recession were allocated randomly to be treated by (GEM 21s) ® with free connective tissue graft (groupI) or GEM 21s with collagen membrane (groupII). Plaque index, bleeding on probing, recession width, recession depth, height of keratinized tissue and digital measurements were recorded at baseline, 1, 3 and 6-months'. Probing pocket depth, clinical attachment level, gingival thickness and Radiographic parameters were recorded at baseline and 6 months'. Root coverage percentage were recorded 6 months postoperative and wound healing index were recorded at 1,3 and 6-months' post-operative .

ELIGIBILITY:
Inclusion Criteria:

* lack of any related medical issues that contraindicate periodontal surgery,
* optimum adherence as confirmed by a positive attitude towards oral hygiene, and successfully showing up for treatment appointments.
* No history of any medications in the previous six months that may interfere with periodontal surgery Gingival thickness for the selected sites should be > 1mm (as measured 2mm apical to gingival margin),
* Clinical attachment level ≥ 4mm measured from cemento-enamel junction till the deepest probing depth.

Exclusion Criteria:

* the presence of class V caries or restoration in the site to be treated,
* previous mucogingival surgery at the selected site.
* Teeth that are tilted, rotated, or have any occlusal abnormalities.
* Smokers and pregnant patients were excluded from the participation.

Ages: 25 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2022-08-30 (Actual); Study Completion 2022-08-30 (Actual)

PRIMARY OUTCOMES:
Recession width | up to 6 months
  the distance between the mesial and distal papillae along the CEJ measured at baseline , 1, 3, and 6 months
recession depth | up to 6 months
  The distance between the CEJ and the gingival margin at the midbuccal aspect of the involved tooth measured at baseline , 1, 3, and 6 months
Height of keratinized tissue | up to 6 months
  distance from the most apical point of the free gingival margin to the mucogingival junction mid-facially measured at baseline , 1, 3, and 6 months
Gingival thickness (Gingival biotype) | up to 6 months
  measured at mid-buccal area 2 mm apical to the free gingival margin measured at baseline, and 6 months postoperatively
radiographic measurements of facial bone level, thickness and density | up to 6 months
  from cone beam CT radiography measured at baseline, and 6 months postoperative
Percentage of root coverage | up to 6 months
  according to the following formula: (RD at baseline - RD at 6 months) / RD at baseline)x100 was calculated after 6 months

SECONDARY OUTCOMES:
probing pocket depth | up to 6 months
  measured from gingival margin to the bottom of the pocket measured at baseline, 3, and 6 months
clinical attachment level | up to 6 months
  measured from CEJ to the bottom of the pocket measured at baseline, 3, and 6 months
Digital measurements | up to 6 months
  all recession areas were photographed The photos were taken by a digital camera at a fixed resolution (mega pixel) taken at baseline, 1,3,and 6 months postoperative
healing index | up to 6 months
  recorded at 1, 3 and 6 months postoperatively (Score 1: uneventful healing while score 3: poor wound healing

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - Malak Mohamed Shoukheba, Tanta
  - Malak Yousef Mohamed Shoukheba, Tanta

IPD SHARING:
Plan to Share IPD: Undecided